CLINICAL TRIAL: NCT05872789
Title: Impact of the Efficacy of Diazepam 1% Oral Gel in Burning Mouth Syndrome
Brief Title: Impact of Diazepam 1% Oral Gel Efficacy in Burning Mouth Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Principal researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-24
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Diazepam; Gels

STUDY DESIGN:
Intervention Model Description: The main objective of this study was to evaluate the efficacy of Diazepam 1% oral gel over placebo in the management of BMS
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diazepam 1% Oral gel (Experimental): Patients were treated with Diazepam 1% oral gel.
  Interventions: Drug: Diazepam 1% oral gel
- Placebo (Placebo Comparator): Patients treated with a placebo gel control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazepam 1% oral gel — Diazepam 1% used with topic oral gel on tongue and palate twice daily.
  Arms: Diazepam 1% Oral gel
Drug: Placebo — Placebo oral gel used on tongue and palate twice daily.
  Arms: Placebo

SUMMARY:
Burning mouth syndrome (BMS) is a syndrome characterized by burning and persistent oral pain, ranging from mild to intense, in the absence of organic disorders of the oral cavity and with a major impact on the quality of life of the sufferer. Although several etiological theories have been proposed to explain BMS, none has been universally accepted to date, and its origin remains unclear. Currently, several scientific evidences would suggest that underlying BMS would be alterations in certain neuropathic mechanisms.

The purpose of the study is to evaluate the efficacy of Diazepam 1% oral gel in the treatment of burning mouth syndrome.

DETAILED DESCRIPTION:
A double-blind placebo-controlled trial is conducted in order to evaluate the efficacy of Diazepam 1% oral gel and determine the statistical significance of the outcome variables. 40 patients with BMS, in two groups:

* case group with Diazepam 1% oral gel (Galenic formulation)
* control group with placebo in oral gel formulation

Follow-up of 2 months

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with BMS who reported a history of continuous oral burning pain for more than 4 months with no clinical signs that could justify the syndrome

Exclusion Criteria:

* • clinically diagnosed with BMS who reported a history of continuous oral burning pain for more than 4 months with clinical signs that could justify the syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Evolution of burning mouth | 2 Months
  Evolution of burning mouth symptoms change through questionnaries. The Visual Pain Analog Scale (VAS) will be used to assess pain, in which the value 0 indicates no pain and the value 100 maximum pain. The Oral Health Impact Profile Short Form (OHIP-14) will be used to assess the impact of oral problems on quality of life, in which the presence or absence of physical pain, functional limitation, psychological distress, physical, psychological and social disabilities, and handicap will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Pubmed